CLINICAL TRIAL: NCT01940445
Title: Impact of Synergistic Sequential Treatment (SST) of Fractional Non-ablative and Q-Switched Lasers on Skin Texture
Brief Title: Impact of Synergistic Sequential Treatment (SST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-M22-13-01
Record Dates: First submitted 2013-09-08; First posted 2013-09-12 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Improvement of Wrinkles/Elastosis as Well as General Skin Tone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ResurFX treatment (Experimental): Fractional Non Ablative (NA) treatment on one side of the face with the M22 ResurFX module
  Interventions: Device: M22 ResurFX
- M22 ResurFX and QS treatment (Experimental): Fractional NA treatment with the M22 ResurFX followed by Q-Switched (QS) laser treatment (SST) on one side of the face
  Interventions: Device: M22 ResurFX and QS

INTERVENTIONS:
Device: M22 ResurFX — Fractional NA treatment (ResurFX) on one side of the face
  Arms: ResurFX treatment
Device: M22 ResurFX and QS — Fractional NA treatment followed by QS laser treatment (SST) on one side of the face
  Arms: M22 ResurFX and QS treatment

SUMMARY:
At least thirty (30) subjects, Fitzpatrick-Goldman Skin Type II-V will be enrolled in 2 clinical sites; each clinic will enroll at least 15 subjects.

Subjects should present visible wrinkles and/or elastosis requiring treatment.

Hypothesis: The SST will improve the appearance of the wrinkles/elastosis as well as general skin tone by at least 25% as compared to M22 ResurFX 1565nm module alone, for at least 75% of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and provide written Informed Consent;
2. Healthy adult, male or female, 30-65 years of age with Fitzpatrick-Goldman skin type II-V;
3. Having suitable facial areas with wrinkles Fitzpatrick-Goldman Wrinkle and Elastosis Score of 3-6 to be treated;
4. Able and willing to comply with the treatment/follow-up schedule and requirements;
5. Women of child-bearing age are required to be using a reliable method of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, Nova ring, partner with vasectomy or abstinence) at least 3 months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

1. Skin type I, VI
2. Pregnant, intending to become pregnant during the course of study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding
3. History of post inflammatory hyperpigmentation
4. Unable or unlikely to refrain from tanning, including the use of tanning booths, during the course of the study
5. Use of photosensitive medication for which light exposure is contraindicated.
6. Use of oral isotretinoin (Accutane®) within 3 months of initial treatment or during the course of the study. Note: skin must regain its normal degree of moisture prior to treatment.
7. Having indurate acne, varicella scars, or severe open wound stages of rosacea.
8. Any dermal/epidermal damage or disorder, mainly vascular or textural lesions, in treated area
9. Prior treatment, such as chemical peel (especially phenol based) or dermabrasion, in treated area within 3 months of initial treatment or during the course of the study;
10. Prior skin laser/light or another device treatment in treated area within 6 months of initial treatment or during the course of the study
11. Prior use of collagen, fat injections or other methods of skin augmentation (enhancement with injected or implanted material) in treated area within 12 months of initial treatment or during the course of the study. Treatment may not be performed at all over permanent dermal implants
12. Prior use of Botox in treatment area within 6 months
13. Prior ablative resurfacing procedure or face lift in treated area with laser or other devices within 12 months of initial treatment or during the course of the study
14. Any other surgery in treated area within 9 months of initial treatment or during the course of the study.
15. Participation in a study of another investigational device or drug involving the same anatomical site within 3 months prior to enrollment or during this evaluation, or if not involving the same anatomical site, as per the Investigator's discretion
16. History of keloid or any other type of hypertrophic scar formation or poor wound healing in a previously injured skin area
17. Showing symptoms of hormonal disorders, as per the Investigator's discretion (such as Melasma, Chloasma)
18. Concurrent inflammatory skin conditions, including, but not limited to, severe rosacea
19. Open laceration or abrasion of any sort on area to be treated during the course of treatment
20. Active Herpes Simplex at the time of treatment or having experienced more than three episodes of Herpes Simplex eruption within a year of study enrollment;
21. Multiple dysplastic nevi in area to be treated
22. Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to treatment (as per the subject's physician discretion)
23. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications
24. Having any form of active cancer at the time of enrollment and during the course of the study or history of skin cancer on the face.
25. Pigmented lesion in the treated area that appears cancerous, pre-cancerous or is not deemed suitable for photo therapy, as determined by a dermatologist.
26. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the anesthesia, treatment, or healing process; Participation in a study of another device or drug within 3 month prior to study enrollment or during this study, and as per the Investigator's discretion, as long as not contradictory to any of the above criteria
27. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse
28. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study.
29. For subjects undergoing test spots: considerable undesired response consisting of skin hypopigmentation (long term whitening), a scar or pre scar formation, or any response deemed by the Investigator as grounds for exclusion.
30. Allergies to anesthetics.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Improvement | 3 months following 3rd treatment
  Investigator subjective evaluation of the extent of wrinkles/elastosis as well as general skin tone improvement of each side of the face at the 3 month follow-up visit as assessed by Fitzpatrick-Goldman Wrinkle Class / Elastosis Score classification and by percentage category scales

SECONDARY OUTCOMES:
Improvement | 1 and 6 months following 3rd treatment
  Investigator subjective evaluation of the extent of wrinkles/elastosis as well as general skin tone improvement of each side of the face at 1 and 6 month follow-up visits as assessed by Fitzpatrick-Goldman Wrinkle Class / Elastosis Score classification and by percentage category scales
Blinded improvement | 1 year following study initiation
  Blinded evaluation of wrinkles and general skin tone improvement at the 1, 3 and 6 months follow-up as compared to baseline using photographs will be performed at the end of the study
Skin response | Following treatments- Baseline, 4, 8 weeks
  Investigator subjective evaluation of skin response following each treatment defined as severity of response and the time it took for it subside for each side of the face
Downtime | Following treatment- baseline, 4, 8 weeks
  Downtime defined as the period of time following the procedure during which the subject felt uncomfortable, unwilling or unable to go out in public due to edema and erythema for each side of the face
Improvement by subject | 1, 3 and 6 months follow up
  Subject subjective opinion of improvement and satisfaction with the treatment based on a percentage category scale for each side of the face
Comfort | Following treatment- baseline, 4, 8 weeks
  Subject subjective assessment of pain and discomfort associated with treatments using a 10 point VAS scale for each side of the face
Biopsies | Immediately post 1st treatment or at 1, 3 or 6 month post last treatment
  Histological analysis of pre auricular tissue samples from both treatment sides with different staining for analysis of changes following treatment
Adverse Events | Following treatment #1, 2 and 3 and all follow up visits
  Safety will be determined by examining the post-treatment occurrences of complications and adverse events throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Girish (Gilly) Munavalli, MD, Principal Investigator — Dermatology, Laser, and Vein Specialists of the Carolinas, PLLC
Locations (1):
- Dermatology, Laser, and Vein Specialists of the Carolinas, PLLC, Charlotte, North Carolina, United States